CLINICAL TRIAL: NCT01431001
Title: Determining Effectiveness of Multi-Coil rTMS for Patients With Major Depressive Disorder: A Pilot Study
Brief Title: Pilot Study in Multi-Coil Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cervel Neurotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS-CPS-TRMD-1
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; MDD; Transcranial Magnetic Stimulation; Depressive Disorder; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coil Configuration A (Experimental): Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator (DSF-rTMS)
  Interventions: Device: Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator (DSF-rTMS)
- Coil Configuration B (Experimental): Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator (DSF-rTMS)
  Interventions: Device: Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator (DSF-rTMS)

INTERVENTIONS:
Device: Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator (DSF-rTMS) — The Cervel Neurotech Deep Shaped-Field repetitive transcranial magnetic stimulator is an investigational rTMS device

SUMMARY:
The purpose of this study is to assess the efficacy of a Deep Shaped-Field repetitive transcranial magnetic stimulation (DSF-rTMS) system in the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder (MDD)
* Mild to moderate level of resistance or intolerance to antidepressant treatment in the current episode.
* Will not become pregnant during study.

Exclusion Criteria:

* Seizure disorder.
* History of brain injury or active CNS disease.
* Metal implants on or in brain, spinal cord, ear, eye or heart.
* Current use of proconvulsant medications (e.g., bupropion).
* Other significant psychiatric disorder.
* Substance use disorder (not including caffeine or nicotine).
* 7 or more failed treatment attempts for depression in one's lifetime.
* Have failed to clinically remit to an adequate trial of ECT or TMS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Remission from depression | baseline through 4 weeks post
  Changes in Hamilton Rating Scale from Depression (HRSD) measured after each block of 5 treatment sessions, 2 weeks post and 4 weeks post

SECONDARY OUTCOMES:
Safety and tolerability of rTMS | baseline through 4 weeks post
  Determined by presence and absence of adverse events recorded daily

CONTACTS AND LOCATIONS:
Overall Officials: AnnaMarie Daniels, Study Chair — Cervel Neurotech
Locations (4):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Rush Medical College, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia